CLINICAL TRIAL: NCT01289964
Title: Randomised Controlled Pilot Study: the Effect of Dry Cupping on Pain and Sensory Thresholds in the Treatment of Chronic Non Specific Neck Pain
Brief Title: The Effect of 5 Times Dry Cupping in the Treatment of Chronic Neck Pain
Acronym: TS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universität Duisburg-Essen (Other)
Responsible Party: Gustav Dobos, University of Duisburg-Essen, Chair of Complementary and Integrative Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DryCupping2009
Record Dates: First submitted 2011-01-31; First posted 2011-02-04 (Estimated); Last update posted 2011-08-19 (Estimated); Status verified 2009-07

CONDITIONS: Neck Pain; Neck Pain Musculoskeletal; Mechanical/Motor Problems With Neck and Trunk
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Waiting list control group (No Intervention): No treatment within the study period, were allowed to continue physiotherapy and medication. Were offered the treatment after finishing the study
- Treatment group (Active Comparator): Received the 5 cupping treatments, application twice a week, non standardised application - individual determinations of trigger points
  Interventions: Procedure: Dry Cupping or fire cupping

INTERVENTIONS:
Procedure: Dry Cupping or fire cupping — 5 dry cupping treatments, application twice a week, non standardised procedure
  Other Names: Cupping is: heating glas cups to create a vacuum on the skin
  Arms: Treatment group

SUMMARY:
The study aims to investigate the influence of 5 dry cupping treatments on chronic non specific neck pain. 50 patients with neck pain are randomised into cupping treatment and waiting list control group at T0 (Day 0). At T1 (Day 7)the investigators evaluate the neck pain (VAS), the neck related disability (NDI), pain related to movement (PRTM) and the quality of life (SF36). To investigate neurophysiological effects of cupping we also measure mechanical detection threshold (MDT), vibration detection threshold (VDT) and pressure pain threshold (PPT) at pain related and control areas. The treatment group then receives 5 cupping treatments over a period of two weeks. After the cupping series resp. a waiting period for the waiting list control group (T2, Day 25) all measurements from T1 are repeated (VAS, NDI, PRTM, SF36, MDT, PPT, VDT). At last, a pain and medication diary is filled in by the patients from T0(Day 0) until T2 (Day 25). The investigators hypothesize, that cupping treatment is effective against neck pain (diary, VAS, NDI, PRTM, SF36) and that it leads to changes on perceptual level (MDT, VDT, PPT), when compared to the waiting list control group.

DETAILED DESCRIPTION:
see above

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 75
* permanent neck pain for at least three months in a row
* a minimum of 40mm of neck pain on a 100mm visual analogue scale (VAS)
* having been in treatment to an orthopaedic or to a neurologist

Exclusion Criteria:

* neck pain caused by trauma, inflammatory or malignant disease, by congenital malformation of the spine or if pain was accompanied by radicular symptoms such as radiating pain, paresis, prickling or tingling.
* invasive treatments within the last 4 weeks, surgery to the spine within the last year, corticosteroid or opioid treatment.
* serious acute or chronic organic disease such as diabetes or cancer, mental disorders, pregnancy, and haemorrhagic tendency or anticoagulation treatment.
* non steroidal pain medication and physiotherapy were allowed if the treatment regimen was not altered for four weeks before and continued during the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2009-07; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Pain intensity | at T2 (Day 25)
  100mm Visual Analogue Scale

SECONDARY OUTCOMES:
pain related to movement | at T2 (Day 25)
  100mm Visual Analogue Scale for 6 movement directions (Irnich, BMJ 2001)
pain diary | from T0 (Day 0) to T2 (Day25)
  Daily rating of pain intensity (numeric rating scale from 0-10)
Neck disability index | at T2 (Day 25)
  NDI measures neck pain complaints (Vernon und Mior 1991)
Quality of Life SF-36 | at T2 (Day 25)
  the sf-36 is a short form health survey consisting of 8 scales to measure functional health and wellbeing (Bullinger & Kirchberger 1998)
mechanical detection threshold MDT | at T2 (Day 25)
  by von Frey filaments to measure perception threshold for light touch (Rolke, Pain, 2006)
vibration detection threshold VDT | at T2 (Day 25)
  with a tuning fork to measure perception threshold for vibration (Rolke, Pain, 2006)
pressure pain threshold PPT | at T2 (Day 25)
  with a pressure gauge algometer to determine threshold for painful pressure (Rolke, Pain, 2006) on the area of maximal neck pain, the adjacent and hand and foot
Side effects | from T1 (Day 7) to T2 (Day 25)
  open question on any side effects or other experiences with the treatment
Medication diary | From T0 (Day 0) to T2 (Day 25)
  patient report used medication during the study period (amount, dose)

CONTACTS AND LOCATIONS:
Overall Officials: Gustav J Dobos, Prof. MD, Principal Investigator — University of Duisburg-Essen, Chair of Complementary and Integrative Medicine
Locations (1):
- Knappschaftskrankenhaus, Essen, North Rhine-Westphalia, Germany

REFERENCES:
- [Result] Lauche R, Cramer H, Choi KE, Rampp T, Saha FJ, Dobos GJ, Musial F. The influence of a series of five dry cupping treatments on pain and mechanical thresholds in patients with chronic non-specific neck pain--a randomised controlled pilot study. BMC Complement Altern Med. 2011 Aug 15;11:63. doi: 10.1186/1472-6882-11-63. PMID 21843336